CLINICAL TRIAL: NCT05339802
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study of the Efficacy and Safety of 9MW1411 Injection Combined With Antibiotics in Patients With Acute Staphylococcus Aureus Skin and Skin Structure Infection
Brief Title: A Phase Ⅱ Clinical Study of 9MW1411 Injection in Acute Bacterial Skin and Skin Structure Infections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW1411-2021-CP201
Record Dates: First submitted 2021-11-16; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Skin Infection
MeSH Terms: conditions — Cellulitis | interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 9MW1411 injection , single administration, intravenous infusion, infusion time 2H (120 ± 15min);
  Interventions: Combination Product: 9MW1411 injection 1 combined with Linezolid
- Cohort 2 (Experimental): 9MW1411 injection , single administration, intravenous infusion, infusion time 2H (120 ± 15min);
  Interventions: Combination Product: 9MW1411 injection 2 combined with Linezolid
- Placebo (Placebo Comparator): 9MW1411 injection placebo, single administration, intravenous infusion, infusion time: 2h (120 ± 15min)
  Interventions: Combination Product: 9MW1411 injection placebo combined with Linezolid

INTERVENTIONS:
Combination Product: 9MW1411 injection 1 combined with Linezolid — After randomization, 9MW1411 injection, single dose, intravenous infusion, linezolid: 600mg, given intravenously or orally every 12 hours, for a total course of treatment not exceeding 14 days.
  Arms: Cohort 1
Combination Product: 9MW1411 injection 2 combined with Linezolid — After randomization, 9MW1411 injection, single dose, intravenous infusion, linezolid: 600mg, given intravenously or orally every 12 hours, for a total course of treatment not exceeding 14 days.
  Arms: Cohort 2
Combination Product: 9MW1411 injection placebo combined with Linezolid — After randomization, 9MW1411 injection placebo, single dose, intravenous infusion, linezolid: 600mg, given intravenously or orally every 12 hours, for a total course of treatment not exceeding 14 days.
  Arms: Placebo

SUMMARY:
In this study, a multicenter, randomized, double-blind, placebo-controlled trial design is used to evaluate the efficacy and safety of two doses of 9MW1411 injection in patients with ABSSSI caused by S. aureus.

The Recommended Phase 2 Dose (RP2D) of 9MW1411 injection for this placebo-controlled study is comprehensively selected based on the results of Phase I clinical trials and preclinical PK/PD analysis. Approximately 90 subjects with ABSSSI caused by S. aureus are planned to be enrolled, and the infection type and presence or absence of single S. aureus infection will be used as randomization stratification factors for all randomized subjects. They are randomized in a 1: 1: 1 ratio.

DETAILED DESCRIPTION:
This study used a multicenter, randomized, double-blind, placebo-controlled trial design to evaluate the efficacy and safety of two doses of 9MW1411 injection in patients with acute staphylococcus aureus skin and skin structure infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 75 years (including 18 and 75 years);
2. One of the following types of skin and skin structure infection is met:

   1. Cellulitis: A diffuse skin infectious disease characterized by diffuse congestion (erythema), edema and/or induration within 7 days of the Screening Visit. The lesion area is at least 75 cm2, calculated as the longest diameter (along the head-to-foot of the human body) multiplied by the widest diameter (perpendicular to the longest diameter), which are measured by the investigator with a ruler.
   2. Wound infection: An infectious disease characterized by purulent drainage from a wound or surgical wound, periwound congestion (erythema), edema and/or induration within 7 days of the Screening Visit. The shortest diameter measured from the perimeter of the wound is at least 5 cm and the lesion area is at least 75 cm2, calculated as the longest diameter (along the head-to-foot of the human body) multiplied by the widest diameter (perpendicular to the longest diameter), which are measured by the investigator with a ruler.
   3. Large cutaneous abscess: An infectious disease characterized by congestion (erythema), edema, and/or induration with collection of pus in the dermis or deeper for the first time within 7 days of the Screening Visit. The shortest diameter measured from the periphery of the abscess is at least 5 cm and the lesion area is at least 75 cm2, calculated as the longest diameter (along the head-to-foot of the human body) multiplied by the widest diameter (perpendicular to the longest diameter), which are measured by the investigator with a ruler.
   4. Burn infection: An infectious disease characterized by purulent drainage with congestion (erythema), edema and/or induration. The shortest diameter measured from the periphery of the burn infection is at least 5 cm and the lesion area is at least 75 cm2 (burn depth is Grade II or higher), calculated as the longest diameter (along the head-to-foot) multiplied by the widest diameter (perpendicular to the longest diameter), which are measured by the investigator with a ruler. Burns occur within 7 days prior to the Screening Visit and cover 10% to 50% of their total body surface area. Patients with burn infections do not exceed 20% of all subjects.
   5. Diabetic foot infection: The subject meets diagnostic criteria for type 1 or 2 diabetes and meets the Infectious Diseases Society of America/International Working Group on Diabetic Foot (IDSA/IWGDF) criteria for moderate infection of diabetic foot (Appendix 1): patients with infection have good systemic function and stable metabolism. However, the patient has ≥ 1 of the following characteristics: ①cellulitis extending > 2 cm around the ulcer, ② lymphatic stripes, ③spreading beneath the superficial fascia, ④deep tissue abscesses; The subject meets the diagnostic criteria for diabetic foot and Wagner grade 2 (Appendix 2) that the ulcer lesion time < 4 weeks: ①If multiple ulcer lesions are present at the same time, the largest lesion is selected as the observed lesion; ②The ulcer lesion is measurable and the lesion area is ≥ 5 cm2, which is calculated as the longest diameter (along the head-foot of the human body) multiplied by the widest diameter (perpendicular to the longest diameter), which are measured by the investigator with a ruler. Patients with diabetic foot infection do not exceed 10% of all subjects.
3. Subjects must have at least two of the following signs/symptoms:

   1. Drainage or discharge of pus;
   2. Erythema;
   3. Fluctuation sensation;
   4. Increased skin temperature;
   5. Edema or induration;
   6. Tenderness;
4. Patients with systemic reactions that meet any of the following:

   1. Fever, defined as oral temperature ≥ 38 °C or axillary temperature ≥ 37.5 °C, or decreased body temperature, i.e., oral temperature < 35 °C or axillary temperature < 34.5 °C;
   2. Peripheral blood white blood cell count ≥ 10 × 109/L or < 4 × 109/L, or neutrophil percentage increased (exceeds the upper limit of the reference value) or banded granulocytes ≥ 15%;
   3. Involvement of lymphatic system: lymphangitis or lymphadenopathy in or adjacent areas of lymphatic drainage at the site of infection;
5. S. aureus infection is judged by any of the following methods prior to randomization:

   1. Rapid diagnostic tests, e.g. FA from BioFire, GX from Cepheid, mass spectrometry, PCR, microarray, second-generation sequencing, etc., are used for preliminary judgement of S. aureus infection. At the same time, the same samples are also used for standard microbial culture without the need to obtain microbial culture results prior to randomization;
   2. Standard microbial culture tests for S. aureus obtained within 72 hours prior to randomization. This sample may be used as a baseline standard microbial culture (including microbial identification, quantitative or semi-quantitative cultures, and susceptibility testing) by each site laboratory.
6. Subjects do not have a fertility plan or sperm donation plan during the study and for 6 months after the end of the study, and voluntarily take effective contraceptive measures:

   1. Female subjects must meet the following conditions: ①non-pregnant or lactating; ②have undergone surgical sterilization or amenorrhea for at least 1 year; ③female subjects of childbearing potential have a negative blood pregnancy test before randomization, and agree to use an effective contraceptive method (e.g., oral contraceptives, condoms, or intrauterine devices) throughout the study or consent to abstinence throughout the study;
   2. Male subjects of childbearing potential agree to use effective barrier contraceptive measures (e.g., condoms) during the study, or their partners agree to use effective contraceptive methods for female subjects as described above, or consent to abstinence throughout the study;
7. Willingness to sign informed consent forms (ICFs);
8. Subjects who can communicate effectively with the investigator, understand and agree to comply with the requirements of this study.

Exclusion Criteria:

1. Patients with uncomplicated skin and skin structure infections, such as furuncles, minor abscesses (no cellulitis/erysipelas around the suppurative area), pustular lesions, superficial or localized cellulitis/erysipelas, and small wound infections (eg, suture abscesses).
2. Patients with confirmed or suspected acute infection of skin and skin structures caused solely by gram-negative bacteria or anaerobes, fungi, and parasites.
3. Presence of any of the following infections:

   Patients with confirmed or suspected osteomyelitis; Patients with confirmed or suspected suppurative arthritis; Patients with implant devices that cannot be removed at the site of infection, such as artificial joints, intravascular catheters, and batteries of permanent pacemakers, etc.; Patients with previous chronic dermatitis or other chronic inflammatory skin lesions, such as eczema and psoriasis, which may affect the judgement of their treatment response; Patients with pressure ulcer infection; Patients with life-threatening infections or infections requiring emergency surgery, such as necrotizing fasciitis, progressive gangrene, and endocarditis, etc.; Patients with infection after human or animal bites (except arthropods).
4. Evidence of any of the following serious immune system disorders:

   Patients with current or expected neutropenia reducing, defined as neutrophil count < 1.5 x 109/L; Patients received cancer chemotherapy, radiotherapy, or strong non-corticosteroid immunosuppressive drugs (e.g., cyclosporine, azathioprine, tacrolimus, immunomodulatory monoclonal antibody therapy, etc.) within the past 3 months; Patients received prednisone at a dose of ≥ 20 mg/day for more than 14 days or an estimated course of treatment more than 14 days prior to enrollment.
5. Patients with known or clinically suspected one or more of the following: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is 3 times higher than the upper limit of normal (ULN); total bilirubin is 2 times higher than the ULN, or evidence of end-stage liver disease (eg, ascites, hepatic encephalopathy).
6. Patients with history or evidence of severe renal disease, or known creatinine clearance (CrCl) < 50 mL/min (estimated using the Cockcroft-Gault formula), or requiring peritoneal dialysis, plasma exchange, hemodialysis, veno-venous dialysis, or other forms of renal filtration.
7. Patients with active or history of autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, etc.) that may relapse, or patients who are at high risks (e.g., organ transplant requiring immunosuppressive therapy).
8. Patients with uncontrolled or uncontrollable hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg), pheochromocytoma, carcinoid syndrome, or hyperthyroidism.
9. Patients with serious or life-threatening condition or organ/system disorders (eg, endocarditis, meningitis, unstable central nervous system disorder, acidosis, or history of lactic acidosis).
10. Patients with burn infection have any of the following: ①Patients with burns of special causes, such as electrical injury, chemical burns, or burns combined with compound injuries (except for arc burns); ②Patients with moderate to severe inhalation injury, severe combined injures, acute respiratory distress syndrome, multiple organ failure, disseminated intravascular coagulation, or acute cardiac insufficiency.
11. Patients with diabetic foot have any of the following: ①Patients with uncontrolled blood glucose (fasting blood glucose > 10 mmol/L) and all types of diabetic coma; ②Patients with canceration at the ulcer site; ③Patients with vascular hypoperfusion of the affected limb, ankle-brachial index (ABI) < 0.6, requiring angioplasty; ④Patients with wound infection with gangrene, which cannot be appropriately cleared by debridement; ⑤The investigator believes that it is likely that a lower knee amputation is necessary.
12. The investigator believes that the subject had any underlying medical conditions affecting participation in the study, including serious heart disease, malignancy, psychosis, ongoing treatment for epilepsy, or a history of untreated epilepsy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Clinical cure in the mITT Population at the Test of cure (TOC) Visit | TOC:Test of cure; 14 days after the last day of linezolid therapy.
  Evaluate the Efficacy of 9MW1411
Incidence and severity of adverse events (AEs)，serious adverse event (SAEs) | From day 1 to day 57（±7） after administration
  Evaluate the Safety of 9MW1411
Incidence of abnormal clinical laboratory findings in 12-lead ECG parameters, vital signs, physical examination | Screening (within 48 hours prior to the first dose of test article) to Follow-up (Day 57±7)
  Evaluate the Safety of 9MW1411
Maximum Observed Concentration (Cmax) | From day 1 to day 57（±7） after administration
  Evaluate the pharmacokinetics profile of 9MW1411
Incidence of anti-drug antibodies | From day 1 to day 57（±7） after administration
  Evaluate the immunogenicity of 9MW1411

SECONDARY OUTCOMES:
Eearly clinical response at 48h~72h after first dose of 9MW1411 | 48h~72h after first dose of 9MW1411
  Evaluate the Efficacy of 9MW1411

OTHER OUTCOMES:
Linezolid Trough Concentration | Before the day of administration, 3 days after administration, 7 days after administration
  To analyze the changing trend of linezolid serum trough concentration in subjects with acute staphylococcus aureus skin and skin structure infection, and to describe the individual differences of linezolid exposure and the correlation between linezolid serum trough concentration and clinical efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Yang NA liecheng, master, Study Director — Mabwell (Shanghai) Bioscience Co., Ltd.
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China